CLINICAL TRIAL: NCT01386424
Title: Screening for LID Clinical Studies Unit Healthy Volunteer Protocols
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110183; 11-I-0183
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-10

CONDITIONS: Zika; Influenza
Keywords: Future; Influenza; Flu; Observation; Vaccine; Healthy Volunteer; HV
MeSH Terms: conditions — Zika Virus Infection; Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers

SUMMARY:
Background:

* The Laboratory of Infectious Diseases (LID) Clinical Studies Unit (CSU) enrolls healthy volunteers into clinical studies to study infectious diseases.
* Viruses can be highly infectious and contagious. They cause considerable illness in the United States each year and a good example of this is influenza (the flu). The LID CSU performs clinical studies to learn about these viral infections and assist in the development of vaccines and treatments for the infections. These clinical studies include influenza "challenge studies" as well as natural history studies and phase I trials involving vaccines for viruses carried by mosquitos such as Zika or Dengue virus.
* In influenza challenge studies studies, doctors expose a person to a flu virus. Then they study the flu through the body's natural healing process. This information will help to find better ways to prevent the flu and may also improve treatments for the flu.
* Natural history studies and phase I trials of new vaccines are performed so the researchers can learn how some viral infections occur and if new vaccines are safe and potentially effective in preventing the infections. In some of these studies, participants experience insect bites with special clean (non-infected) insects (such as mosquitos) to better understand the role of insects in these infections.

Objectives:

- To screen healthy volunteers for future CSU studies.

Eligibility:

- Healthy people between the ages of 18 and 65

Design:

* The 3- to 5-hour screening exam includes the following:
* Medical history and physical exam
* Standard blood tests including pregnancy, Hepatitis B and C, and HIV tests
* Standard urine drug testing
* Electrocardiogram (ECG) to test heart rhythm and function
* Chest x-ray
* Eligible volunteers are enrolled in the study for up to 1 year, until they take part in a CSU study or are found to be ineligible to participate.
* Volunteers may withdraw from the study pool at any time.

DETAILED DESCRIPTION:
The high morbidity and mortality associated with both pandemic and seasonal influenza and the anticipation for future influenza pandemics puts influenza front and center in infectious disease research. Because the natural history and pathogenesis of human influenza has not been well characterized and cannot be adequately studied in animal models or with current in vitro techniques, important questions about influenza pathogenesis can only be approached through human challenge studies.

Previous human challenge studies have addressed some aspects of the natural history by evaluating the timing of viral replication, shedding, clinical symptoms, and innate and adaptive immune responses. Although these studies have provided important information, all but one was performed prior to 1990. Without exception, these studies had limitations due to the scope of the study and/or the scientific techniques available at that time.

While initially the protocol was designed to screen participants for influenza challenge studies, we have expanded our scope of research to include emerging and re-emerging infectious diseases.The primary goal of this study is to collect and store serum and RNA samples and obtain clinical and laboratory data from volunteers to determine in advance if they are potentially eligible to participate in future clinical studies. To accomplish this objective, up to 5000 participants will be enrolled in this protocol at the NIH Clinical Center clinic or day hospital in order to maintain a pool of participants who have been evaluated and can be screened for future LID Clinical Studies Unit protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Greater than or equal to 18 and less than or equal to 65 years old, and have no significant health abnormalities
  2. Willing to consider taking part in a future LID Clinical Studies Unit healthy volunteer study
  3. A female participant is eligible for this study if she is any of the following:
* Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are post-menopausal, as defined by no menses in greater than or equal to 1 year)
* Of childbearing potential but agrees to practice effective contraception or abstinence (from heterosexual sex) for 4 weeks prior to enrolling into a spceific study and during the study.

NOTE: Acceptable methods of contraception may include one or more of the following: 1) male partner who is sterile prior to the female participant's entry into the study and is the sole sexual partner for the female participant; 2) implants of levonorgestrel; 3) injectable progestogen;, 4) an intrauterine device with a documented failure rate of less than 1percent; 5) oral contraceptives; or 6) double barrier methods including diaphragm or condom with a spermicide.

4. Willing to have samples stored for future research

EXCLUSION CRITERIA:

1. Self-reported history of any significant medical condition including but not limited to:

   * Chronic pulmonary disease (such as asthma, emphysema)
   * Chronic cardiovascular disease (cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects)
   * Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (diabetes mellitus, renal dysfunction, hemoglobinopathies)
   * Immunosuppression or cancer
   * Neurological and neuro-developmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures)
   * Drug and/or alcohol dependency and/or abuse
2. Any condition that, in the judgment of the Principal Investigator, is a contraindication to protocol participation or impairs the volunteer s ability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Population
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-07-20 (Actual)

PRIMARY OUTCOMES:
Find Healthy volunteers for research | One time for a participant, 20 year open study
  The primary goal of this study is to collect and store serum and RNAsamples and obtain clinical and laboratory data from volunteers todetermine in advance if they are potentially eligible to participate infuture LID Clincal Studies Unit protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Carrat F, Vergu E, Ferguson NM, Lemaitre M, Cauchemez S, Leach S, Valleron AJ. Time lines of infection and disease in human influenza: a review of volunteer challenge studies. Am J Epidemiol. 2008 Apr 1;167(7):775-85. doi: 10.1093/aje/kwm375. Epub 2008 Jan 29. PMID 18230677
- [Background] Brown TA, Murphy BR, Radl J, Haaijman JJ, Mestecky J. Subclass distribution and molecular form of immunoglobulin A hemagglutinin antibodies in sera and nasal secretions after experimental secondary infection with influenza A virus in humans. J Clin Microbiol. 1985 Aug;22(2):259-64. doi: 10.1128/jcm.22.2.259-264.1985. PMID 4031039
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-I-0183.html